CLINICAL TRIAL: NCT02260206
Title: Impact of Colchicine Therapy on Arrhythmia Recurrence After Acute Pericardial Effusion Following Catheter Ablation of Atrial Fibrillation
Brief Title: Impact of Colchicine Therapy on Arrhythmia Recurrence After Acute Pericardial Effusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, MD, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: colchicine
Record Dates: First submitted 2014-10-05; First posted 2014-10-09 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pericardial Effusion
Keywords: Pericardial Effusion; Colchicine; arrhythmia Recurrence; pericardiocentesis
MeSH Terms: conditions — Pericardial Effusion | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: None (Open label)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine (Experimental): Impact of Colchicine therapy on arrhythmia Recurrence after Acute Pericardial Effusion following Catheter Ablation of Atrial Fibrillation
  Interventions: Drug: Colchicine
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Colchicine — Impact of Colchicine therapy on arrhythmia Recurrence after Acute Pericardial Effusion following Catheter Ablation of Atrial Fibrillation
  Other Names: Impact of Colchicine
  Arms: Colchicine

SUMMARY:
The effects colchicine administration for acute pericardial effusion after radiofrequency catheter ablation (RFCA) of atrial fibrillation on the recurrences of arrhythmia.

DETAILED DESCRIPTION:
RFCA was started as a rhythm control of atrial fibrillation about 10 years before and the superiority of RFCA to medical treatment has been continuously reporting, so RFCA is globally performed nowadays. Acute pericardial effusion could occur during RFCA as complication, that might be developed to cardiac tamponade needed immediate pericardiocentesis. The inflammation developed after pericardiocentesis might be associated with the recurrences of atrial fibrillation, it could be presumed by the frequent occurrence of atrial fibrillation after open-heart surgery. The inflammation can be suppressed by administration of colchicine and the effects of colchicine have been proven to decrease the development of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients needed to pericardiocentesis during RFCA for paroxysmal or persistent atrial fibrillation.

Exclusion Criteria:

* Hypersensitivity on Colchicine
* The existence of intra-cardiac thrombus on trans-esophageal echocardiography
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2019-09 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
recurrence of atrial arrhythimia | 1 year after colchicines administration
  Assessment of the recurrence of atrial arrhythimia 1 year after colchicines administration

SECONDARY OUTCOMES:
recurrence of atrial arrhythimia | 3 year after colchicines administration
  Assessment of the recurrence of atrial arrhythimia 3 year after colchicines administration

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seog Oh, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Cho Gu, South Korea

IPD SHARING:
Plan to Share IPD: No